CLINICAL TRIAL: NCT04551027
Title: Assessing the Effect of Compensatory Cognitive Intervention for Functional Capacity, Cognitive Functions and Severity of Symptoms Among People With Severe Mental Illness
Brief Title: Assessing the Effect of Compensatory Cognitive Intervention Among People With Severe Mental Illness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, ido lurie, Director of adult clinic, Shalvata Mental Health Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0003-20-SHA
Record Dates: First submitted 2020-08-14; First posted 2020-09-16 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Mood Disorders; Schizophrenia; Schizoaffective Disorder
Keywords: compensatory cognitive treatment; mental illness; cognitive strategies; everyday functioning
MeSH Terms: conditions — Mood Disorders; Schizophrenia; Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- compensatory cognitive treatment (Experimental): compensatory cognitive treatment intervention, focusing on learning cognitive strategies to overcome cognitive deficits.
  Interventions: Behavioral: compensatory cognitive treatment
- control group (No Intervention): standard ambulatory treatment

INTERVENTIONS:
Behavioral: compensatory cognitive treatment — a brief group compensatory cognitive intervention including 12 meetings of 1 hour in a group of five and focuses on these cognitive domains: prospective memory, vigilance and attention, memory and learning and executive functions
  Arms: compensatory cognitive treatment

SUMMARY:
The aim of this study is to assess the efficacy of a short term compensatory cognitive group intervention - the Compensatory Cognitive Training (CCT) among people with severe mental illnesses, receiving ambulatory treatment

DETAILED DESCRIPTION:
This study includes two experimental arms to research cognitive compensatory group treatment in severe mental illness population. The study consists of 4 primary phases: recruitment, assessment, intervention and post-intervention assessment. Two arms involve an ambulatory participants. participants are assigned to an intervention or control group according to the order of recruitment. Assessment and post-assessment phases include assessments of functional capacity, cognitive functions and severity of symptoms.

Intervention includes 12 group sessions in a small group of five participants, focusing on learning compensatory strategies aimed to improve attention, concentration, learning, memory, organization, and problem-solving in order to improve everyday functioning. Interventions will be performed in addition to standard ambulatory treatment. The control group will receive standard ambulatory treatment only.

ELIGIBILITY:
Inclusion Criteria:

* basic knowledge in Hebrew
* diagnosed according to the ICD -10 with severe mental illness: schizophrenia, bipolar disease, schizoaffective disorder or major depression
* Patients are treated with neuroleptic medication for at least four weeks.

Exclusion Criteria:

* acquired neurological disorders including dementia and brain injury.
* Developmental neurological disorders including developmental intellectual disability and autistic spectrum disorders.
* Regular Electro convulsive therapy treatment with frequency of twice a month or more.
* People to whom a guardian has been appointed
* Current addiction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline functional capacity at 12 weeks : The Observed Tasks of Daily Living-Revised (OTDL-R) | 30 min duration at week 0 ; week 12
  OTDL-R is an objective, performance-based evaluation of the subjects' ability to perform daily life activities in the following areas: Medication management, communication and finances management. The final score ranges from 0 (not independent) to 28 (independent).

SECONDARY OUTCOMES:
Change from baseline cognitive functions at 12 weeks: The Cognitive Problems and Strategies Assessment (CPSA) | 10 min at week 0 ; week 12
  CPSA is a self-reported questionnaire on personal experience of cognitive difficulties and usage of cognitive strategies. The final score for each scale ranges from 0 (Rarely/ Never) to 3 (always)
Change from baseline severity of clinical symptoms at 12 weeks: Clinical Global Impression (CGI) | week 0 ; week 12
  a scale used by the clinician to assess the severity of symptoms according to symptoms, behaviour and function in the last week. The final score ranges from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients)
Change from baseline cognitive functions at 12 weeks: The Neurobehavioral Cognitive Status Examination (COGNISTAT) | 20 min at week 0 ; week 12
  COGNISTAT is a cognitive screening test for 3 basic cognitive functions: Orientation, Attention, Memory Registration and 5 major cognitive functions: Language (Comprehension, Repetition, Naming), Constructional Ability, Memory, Calculation Skills, Executive Skills (Reasoning, Judgment). The final scores for the subtests ranges from 0 (severe impairment) to 4, 6, 8 or 12 (average range)
Change from baseline cognitive functions at 12 weeks: Rey- Ostereich Complex Figure | 20 min at week 0 ; week 12
  a cognitive performance test evaluating instant visual memory and visual organization. The final score for accuracy ranges from 0-36 as higher score indicate better accuracy. The final score for the general performance of the task ranges from 1 (very reasonable) to 7 (not at all reasonable).
Change from baseline cognitive functions at 12 weeks: Trail Making Test A & B (TMT) | 3 min at week 0 ; week 12
  Paper and pencil neuropsychological test that evaluating processing speed and shifting. The final score represents the time length in which the subject completed the test.
Change from baseline cognitive functions at 12 weeks: Behavioral Assessment of the Dysexecutive Syndrome (BADS): key searching test | 1 min at week 0 ; week 12
  a cognitive performance test evaluating problem solving, regulating and monitoring behavior. The final score ranges from 0-4, Higher score is a better result.
Change from baseline cognitive functions at 12 weeks: Category Fluency Test (CFT) | 1 min at week 0 ; week 12
  A neuropsychological test evaluating the ability to retrieve information from memory in a limited amount of time. The final score represents the number of words the subject succeeded to retrieve in the limited time. Higher score is a better result.

CONTACTS AND LOCATIONS:
Overall Officials: Ido Lurie, M.D, Principal Investigator — Director of Adult clinic, Shalvata Mental Health Center; Lena Lipskaya, P.H.D, Study Director — The Department of Occupational Therapy, The Stanley Steyer School of Health Professions, Sackler Faculty of Medicine,Tel Aviv University
Locations (1):
- Shalvata mental health center, Hod HaSharon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Twamley EW, Burton CZ, Vella L. Compensatory cognitive training for psychosis: who benefits? Who stays in treatment? Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S55-62. doi: 10.1093/schbul/sbr059. PMID 21860048
- [Background] Twamley EW, Savla GN, Zurhellen CH, Heaton RK, Jeste DV. Development and Pilot Testing of a Novel Compensatory Cognitive Training Intervention for People with Psychosis. Am J Psychiatr Rehabil. 2008 Apr;11(2):144-163. doi: 10.1080/15487760801963678. PMID 19198664
- [Background] Twamley EW, Thomas KR, Burton CZ, Vella L, Jeste DV, Heaton RK, McGurk SR. Compensatory cognitive training for people with severe mental illnesses in supported employment: A randomized controlled trial. Schizophr Res. 2019 Jan;203:41-48. doi: 10.1016/j.schres.2017.08.005. Epub 2017 Aug 18. PMID 28823720
- [Background] Twamley EW, Vella L, Burton CZ, Heaton RK, Jeste DV. Compensatory cognitive training for psychosis: effects in a randomized controlled trial. J Clin Psychiatry. 2012 Sep;73(9):1212-9. doi: 10.4088/JCP.12m07686. Epub 2012 Aug 7. PMID 22939029
- See also: A website which gives free access to the manuals of the CCT intervention — http://www.cogsmart.com/